CLINICAL TRIAL: NCT02424435
Title: Open-label Pilot Study of Methylprednisolone for the Treatment of Patients With Friedreich Ataxia (FRDA)
Brief Title: Methylprednisolone Treatment of Friedreich Ataxia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Friedreich's Ataxia Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-011801
Record Dates: First submitted 2015-04-16; First posted 2015-04-23 (Estimated); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Friedreich Ataxia
Keywords: Friedreich Ataxia; FRDA
MeSH Terms: conditions — Friedreich Ataxia | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Methylprednisolone (Experimental): This is an open-label study of methylprednisolone in patients with FRDA. Subjects will begin oral administration of 48 mg methylprednisolone at day 1 and will decrease their administered dose by 8 mg per day. After 6 days, subjects will spend 22 days off medication before repeating the same treatment cycle. Last dosing cycle of methylprednisolone will be administered at 24 weeks after baseline. Visits will occur at weeks 2, 6, 14, 26, and 30 following baseline.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — Oral tablets of methylprednisolone 8 mg. Subjects will receive a monthly prescription bottle of 25 tablets (standard quantity) and will self-administer 21 tablets over a 28-day dosing cycle.

SUMMARY:
This study will explore whether methylprednisolone treatment is safe, well-tolerated, and beneficial in patients that are diagnosed with Friedreich Ataxia (FRDA). The study will also explore if methylprednisolone has any effects on biomarkers associated with FRDA. All subjects in the study will receive the same steroid treatment.

DETAILED DESCRIPTION:
Context:

Friedreich ataxia (FRDA) is a progressive neurodegenerative disease of children and adults for which there is presently no therapy. One of the hallmarks of FRDA is a deficiency of frataxin protein, causing dysregulation of iron metabolism, lack of detoxification, and increased iron bioavailability. The accumulation of iron in mitochondria leads to increased sensitivity to oxidative stress. A secondary inflammatory response has also been proposed to be present in FRDA, as revealed in autopsy studies and in the alteration of immune pathways in microarray analysis. Inflammation in FRDA raises the possibility of a therapeutic benefit from anti-inflammatory steroid treatment, as inflammation may directly underlie multiple complications of FRDA including cardiomyopathy. In support of this theory are clinical observations and patient self-reports of improvement of ataxia symptoms following the prescription of steroids for indications other than the primary FRDA diagnosis.

Objectives:

Primary: To assess the effect of oral administration of methylprednisolone on the functional performance scores of patients with FRDA using the Timed 25-Foot Walk (T25FW).

Secondary: To assess the effect of methylprednisolone on neurological performance measures (Friedreich Ataxia Rating Scale, 9-Hole Peg Test, 1-minute walk, home-based measures of gait, hand function and speech assessed through smartphone application) and to assess the safety and tolerability of methylprednisolone in the FRDA population.

Study Design:

This study is an open-label clinical trial of methylprednisolone in patients with FRDA.

Setting/Participants:

This study will take place at the Children's Hospital of Philadelphia as an outpatient trial in 5 children who are at least 5 years and less than 10 years of age, and in 5 adults ages 45 years and older, with genetically confirmed FRDA.

See below for description of study intervention and measures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with FRDA confirmed by genetic testing who are able to walk 25 feet (assistive devices allowed).
* Children between ages 5 and less than 10 years or adults ages 45 years and older at screening.
* Stable doses of all medications, vitamins and supplements for 30 days prior to study entry and for the duration of the study. Throughout the study, all possible efforts will be made to maintain stable doses of concomitant medications.
* Females who are not pregnant or breast feeding, and who do not intend to become pregnant. Females of child-bearing potential must use a reliable method of contraception and must provide a negative urine pregnancy test at screening.
* Informed consent for adult participants, parent/guardian permission (informed consent) and child assent for pediatric participants.

Exclusion Criteria:

* Patients unable to walk 25 feet.
* Treatment with methylprednisolone or cyclic methylprednisolone during the 3 previous months before inclusion.
* Treatment with gamma interferon, immunoglobulin G or other immunomodulating treatment the 3 previous month before inclusion
* Immunosuppressive treatment within 6 month of inclusion
* Prior history of a disease associated with immune dysfunction
* Poorly controlled Diabetes Mellitus (HbA1C > 9.0)
* History of untreated or uncontrolled hypertension
* Presence of infectious disease or other active infections which the treating physician finds relevant
* Active or previous history of liver or renal failure
* Known history of renal insufficiency or creatinine > 2 x upper limit of normal (ULN)
* Active infection at time of screening
* History of known osteoporosis

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change in the Timed 25 Foot Walk (T25FW) Score | This outcome will be measured at baseline and 26 weeks
  The T25FW is a quantitative mobility and leg function performance test based on a timed 25-foot walk. The subject is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible. The time is calculated from the initiation of the instruction to start and ends when the subject has reached the 25-foot mark. The task is immediately administered again by having the subject walk back the same distance. Subjects may use assistive devices when doing this task.

SECONDARY OUTCOMES:
Change in the Friedreich Ataxia Rating Scale (FARS) Score | This outcome will be measured at baseline and 26 weeks
  The Friedreich Ataxia Rating Scale (FARS) is neurological rating scale specifically developed and validated for FRDA. The FARS includes assessments of stance, gait, upper and lower limb coordination, speech, proprioception and strength. In addition to the standard neurological examination, the FARS contains three quantitative performance measures and a component that assesses activities of daily living (ADL). Quantitative performance measures include the nine-hole peg test, and a timed 25-foot walk. FARS scores correlate significantly with functional disability, activities of daily living scores and disease duration. The scores from the three subscales are added to generate a total score ranging from 0 to 159, with a higher score indicating a greater level of disability.
Change in The 1-Minute Walk Distance | This outcome will be measured at baseline and 26 weeks
  The 1-Minute Walk is a quantitative mobility and leg function performance test based on distance traveled in 1 minute. The subject is directed to one end of a clearly marked 25-foot course and instructed to walk back and forth as quickly as possible for 1 minute. The distance is calculated by measuring how far the subject travels along the 25-foot course. Subjects may use assistive devices during this task.
Change in the Change in the 9-Hole Peg Test (9HPT) Time | This outcome will be measured at baseline and 26 weeks
  The 9HPT is a brief, standardized, quantitative test of upper extremity function. Both the dominant and non-dominant hands are tested twice. The subject is seated at a table with a small, shallow container holding nine pegs and a wood or plastic block containing nine empty holes. The total time to complete each of four trials is recorded. Two consecutive trials with the dominant hand are immediately followed by two consecutive trials with the non-dominant hand.

CONTACTS AND LOCATIONS:
Overall Officials: David R Lynch, MD PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States